CLINICAL TRIAL: NCT02181036
Title: Effects of Family Work Shop for Children With Speech Developmental Delays
Brief Title: Effects of Work Shop for Children With Developmental Delays
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DOH-SKH-103-07
Record Dates: First submitted 2014-06-30; First posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Developmental Delays
Keywords: Family work shop; speech developmental delays; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- family work shop (Experimental): 2 to 3 hours per session, one session per week, for a total of 6 weeks of family work shop
  Interventions: Other: family work shop

INTERVENTIONS:
Other: family work shop — 2-3 hours per session, one session per week, a total of 6 weeks of family work shop

SUMMARY:
To identify the effects of family work shop for children with speech developmental delays.

DETAILED DESCRIPTION:
To assess the improvement of functional performance of children with speech developmental delays by 2-3 hours per session, one session per week, a total of 6 weeks of family work shop

ELIGIBILITY:
Inclusion Criteria:

* 18 M/O to 36 M/O of children with speech development delay

Exclusion Criteria:

* less than 18 M/O older than 36 M/O

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
changes of pediatric health related quality of life (Pediatric Quality of Life Inventory) | participants will be evaluated at before and after 6 weeks of work shop
  participants receive one 2-hour session of work shop per week for a 6-week duration

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Study Director — Taipei Medical University
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan